CLINICAL TRIAL: NCT06515665
Title: Investigation of the Effectiveness of Diabetic Recovery Shoes and Artificial Intelligence Supported Structured Exercise Program in Individuals with Diabetic Foot Receiving Hyperbaric Oxygen Therapy
Brief Title: Effectiveness of Diabetic Recovery Shoes and Artificial Intelligence Supported Structured Exercise Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Tezel Yıldırım Şahan, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Effectiveness of Recovery Shoe
Record Dates: First submitted 2024-05-13; First posted 2024-07-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: diabetic foot ulcer; foot orthoses; artificial intelligence
MeSH Terms: conditions — Diabetic Foot | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: There are 3 groups. Fisrt group has therapeutic foot orthosis. Second group has orthosis and exercises with artificial intelligence. Third group is control group.
Who Masked: Participant
Masking Description: A online site named "randomizer.org " gave us a random queue. Participant do not know their queue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- therapeutic foot orthosis (Active Comparator): foot orthosis will be applied to this group of participants. For 6 weeks they will be asked to use these foot orthoses. Before and after evaluations will be repeated.
  Interventions: Behavioral: therapeutic foot orthosis
- exercises (Active Comparator): this group of participants will be exercised with foot orthoses accompanied by artificial intelligence. For 6 weeks, they will be asked to use these foot orthoses and do their exercises. Before and after evaluations will be repeated.
  Interventions: Behavioral: therapeutic foot orthosis
- control (Active Comparator): this group of participants will be assessed at the beginning and end of the 6 weeks without any intervention.
  Interventions: Behavioral: therapeutic foot orthosis

INTERVENTIONS:
Behavioral: therapeutic foot orthosis — They will be asked to behaviorally wear this shoe and perform the exercises daily for 6 weeks.
  Other Names: exercises

SUMMARY:
This study aims to evaluate the effectiveness of the diabetic recovery sandal and artificial intelligence supported structured exercise program in individuals diagnosed with diabetic foot receiving hyperbaric oxygen therapy. The study will include 66 individuals between the ages of 40-65 who have received a diagnosis of diabetic foot from a specialist doctor, have a forefoot wound and receive hyperbaric oxygen therapy. The included individuals will be randomly divided into 3 groups. All participants will be provided with appropriate wound care and dressing and will be randomly divided into 3 groups. Artificial intelligence assisted exercise (exercise group) will be applied to the 1st group. Group 2 will receive artificial intelligence-assisted exercises and healing sandals. For 6 weeks, diabetic foot exercises and diabetic recovery sandal use will be provided (Exercise + sandal group). 3 groups will not receive any contribution (Control group). Balance, performance, wound healing and muscle strength evaluations will be performed before and after the application. Balance assessments will be evaluated by timed get up and walk test, performance by 1 min walk test, wound healing by Imitto measure phone application and muscle strength assessments by manual muscle tests.Awareness of the use of recovery sandals, hyperbaric oxygen therapy and foot exercises will be increased. Attention will be drawn to the creation of new education programs for people with low education or perception, and necessary measures will be taken in cases where risk is identified. In addition, early detection of recurrent ulcers or amputations in individuals who may increase the level of amputation will increase the risk of hospitalization and at the same time increase the cost of care that needs to be spent during hospitalization.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of the diabetic recovery sandal and artificial intelligence supported structured exercise program in individuals diagnosed with diabetic foot receiving hyperbaric oxygen therapy. The study will include 66 individuals between the ages of 40-65 who have received a diagnosis of diabetic foot from a specialist doctor, have a forefoot wound and receive hyperbaric oxygen therapy. The included individuals will be randomly divided into 3 groups. All participants will be provided with appropriate wound care and dressing and will be randomly divided into 3 groups. Artificial intelligence assisted exercise (exercise group) will be applied to the 1st group. Group 2 will receive artificial intelligence-assisted exercises and healing sandals. For 6 weeks, diabetic foot exercises and diabetic recovery sandal use will be provided (Exercise + sandal group). 3 groups will not receive any contribution (Control group). Balance, performance, wound healing and muscle strength evaluations will be performed before and after the application. Balance assessments will be evaluated by timed get up and walk test, performance by 1 min walk test, wound healing by Imitto measure phone application and muscle strength assessments by manual muscle tests.Awareness of the use of recovery sandals, hyperbaric oxygen therapy and foot exercises will be increased. Attention will be drawn to the creation of new education programs for people with low education or perception, and necessary measures will be taken in cases where risk is identified. In addition, early detection of recurrent ulcers or amputations in individuals who may increase the level of amputation will increase the risk of hospitalization and at the same time increase the cost of care that needs to be spent during hospitalization. It is also expected to provide evidence to health professionals working in this field.

ELIGIBILITY:
Inclusion Criteria:

* individuals were ability to walk 10 meters with a maximum of one support,
* at most one amputated toe, no thumb,
* accessible to electronic devices with internet,
* no vision and hearing problems,
* no problems that may affect cooperation,
* receiving Hyperbaric Oxygen Therapy.

Exclusion Criteria:

* having major amputations,
* having an orthopedic or other neurological problem,
* having a congenital disability,
* having proximal lower extremity,
* amputation excluding the finger,
* having bilateral finger amputation.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Balance Evaluation of Individuals with Diabetic foot | Before and after 6 week
  time up and go test
Performance Evaluation of Individulas With Diabetic Foot | before and after 6 week
  one minute walk test
Wound Healing Evaluation of Individulas With Diabetic Foot | before and after 6 week
  Photos will be taken with a phone application called Imit measure.

SECONDARY OUTCOMES:
Comparing the effectiveness of the diabetic recovery orthosis and exercises on balance | before and after 6 week
  Comparing week six assessments
Comparing the effectiveness of the diabetic recovery orthosis and exercises on performance | before and after 6 week
  Comparing week six assessments
Comparing the effectiveness of the diabetic recovery orthosis and exercises on wound healing | before and after 6 week
  Comparing week six assessments

CONTACTS AND LOCATIONS:
Overall Officials: Tezel Y Şahan, phD, Study Chair — University of Health science
Locations (1):
- University of Health Science, Ankara, Kecıoren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
will be decided after the study is finished.

REFERENCES:
- [Background] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678
- [Background] Buldt AK, Menz HB. Incorrectly fitted footwear, foot pain and foot disorders: a systematic search and narrative review of the literature. J Foot Ankle Res. 2018 Jul 28;11:43. doi: 10.1186/s13047-018-0284-z. eCollection 2018. PMID 30065787
- [Background] Collings R, Freeman J, Latour JM, Paton J. Footwear and insole design features for offloading the diabetic at risk foot-A systematic review and meta-analyses. Endocrinol Diabetes Metab. 2020 Apr 11;4(1):e00132. doi: 10.1002/edm2.132. eCollection 2021 Jan. PMID 33532602
- [Background] Ercan E, Aydin G, Erdogan B, Ozcelik F. The effect of hyperbaric oxygen therapy on hematological indices and biochemical parameters in patients with diabetic foot. Medicine (Baltimore). 2024 Mar 22;103(12):e37493. doi: 10.1097/MD.0000000000037493. PMID 38518039